CLINICAL TRIAL: NCT03574792
Title: A Randomized, Open-Label Study to Assess the Pain, Toxicity, and Quality of Life Effects of Adding Venlafaxine to the Pain Management Regimen for Patients Treated With Chemoradiation for Head and Neck Cancer
Brief Title: Gabapentin, Methadone, and Oxycodone With or Without Venlafaxine Hydrochloride in Managing Pain in Participants With Stage II-IV Squamous Cell Head and Neck Cancer Undergoing Chemoradiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 61117; NCI-2018-01055 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 61117 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2018-06-11; First posted 2018-07-02 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8
MeSH Terms: interventions — Gabapentin; Methadone; Oxycodone; Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (gabapentin, methadone, oxycodone) (Active Comparator): Participants receive gabapentin PO daily or TID. Participants may also receive methadone PO TID and oxycodone PO every 8 hours as needed. Treatment continues for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gabapentin; Drug: Methadone; Drug: Oxycodone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (gabapentin, methadone, oxycodone, venlafaxine) (Experimental): Participants receive gabapentin, methadone, and oxycodone as in Arm I and venlafaxine PO BID or venlafaxine hydrochloride extended release daily for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gabapentin; Drug: Methadone; Drug: Oxycodone; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Venlafaxine; Drug: Venlafaxine Hydrochloride Extended Release

INTERVENTIONS:
Drug: Gabapentin — Given PO
  Other Names: Gralise; Neurontin
Drug: Methadone — Given PO
Drug: Oxycodone — Given PO
  Other Names: Oxycodone SR
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Venlafaxine — Given PO
  Arms: Arm II (gabapentin, methadone, oxycodone, venlafaxine)
Drug: Venlafaxine Hydrochloride Extended Release — Given PO
  Other Names: Effexor XR; Venlafaxine HCl ER
  Arms: Arm II (gabapentin, methadone, oxycodone, venlafaxine)

SUMMARY:
This trial studies how well gabapentin, methadone, and oxycodone with or without venlafaxine hydrochloride work in managing pain in participants with stage II-IV squamous cell head and neck cancer undergoing chemoradiation therapy. Gabapentin may reduce the need for these pain medications if given at the start of radiation therapy. Methadone and oxycodone may help relieve pain caused by cancer. Venlafaxine hydrochloride may prevent or improve pain caused by cancer. It is now yet known whether giving gabapentin, methadone, and oxycodone with venlafaxine hydrochloride will work better in managing pain in participants with squamous cell head and neck cancer undergoing chemoradiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the pain-reduction effects of adding venlafaxine to a regimen of gabapentin and methadone to control pain during and after chemoradiation.

SECONDARY OBJECTIVES:

I. To assess the effect of venlafaxine hydrochloride (venlafaxine) of the rate of toxicities possibly or probably related to the pain control regimen.

TERTIARY OBJECTIVES:

I. The effect of venlafaxine on other quality of life scores, patient nutrition, hydration status, and opioid requirements during and after chemoradiotherapy (CRT).

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants receive gabapentin orally (PO) daily or 3 times a day (TID). Participants may also receive methadone PO TID and oxycodone PO every 8 hours as needed. Treatment continues for up to 12 months in the absence of disease progression or unacceptable toxicity.

ARM II: Participants receive gabapentin, methadone, and oxycodone as in Arm I and venlafaxine PO twice daily (BID) or venlafaxine hydrochloride extended release daily for up to 12 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up at 4 weeks, 3, 6, 9, and 12 months, and then every 6 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for chemoradiation therapy of the head and neck.
* Patients must have adequate renal function to undergo platinum based chemotherapy. This will mean a baseline creatinine level (Cr) no greater than 1.5 times the upper limit of normal.
* Have a pathologic diagnosis of squamous cell carcinoma of the head and neck region
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2.
* Ability to swallow and/or retain oral or per tube medication.
* Patients of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Patients who have previously been treated with surgery or radiation for head and neck cancer and/or are being treated for recurrent head and neck cancer.
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Any patients prescribed medications for chronic and/or long term pain and/or neuropathy will be excluded, including patients under treatment of a pain specialist or substance-abuse programs. Acute post-op medications are allowed if the patient has discontinued them prior to initiating study.
* Any patients prescribed a selective serotonin reuptake inhibitor (SSRI), serotonin and norepinephrine reuptake inhibitor (SNRI), tricyclic antidepressant (TCA), monoamine oxidase inhibitors (MAOIs), dextromethorphan, triptan, tryptophan supplements, IV methylene blue, linezolid or any other medication that may increase risk of serotonin syndrome, as deemed by the investigator?s opinion.
* Any patients with suspected or known, current or recent (within last 5 years) use of cocaine, amphetamines, lysergic acid diethylamide (LSD), 3,4- methylenedioxymethamphetamine (MDMA), or any other drug of abuse that may increase risk of serotonin syndrome, as deemed by the Investigator?s opinion.
* Any patients with history of suicide-related events, or those exhibiting a significant degree of suicidal ideation.
* Patients with acute narrow-angle glaucoma.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing female patients.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator?s opinion deems the patient an unsuitable candidate to receive study drug.
* Received an investigational agent within 30 days prior to enrollment.
* Patients on dialysis or with transplanted organs.
* Patients already enrolled on other studies of systemic pain control agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Participant pain levels per European Organization for Research and Treatment of Cancer (EORTC) Head and Neck Cancer Module (EORTC QLQ-H and N35) | Up to 24 months
  Change in Pain Scale score is measured repeatedly during the 7-week radiation treatment process, and periodically for as long as the patient receives pain management treatment, up to 24 months after enrollment. The magnitude, direction and 95% confidence interval for the adjusted interaction term estimate will be used to describe the effect venlafaxine in improving the pain management regimen.

SECONDARY OUTCOMES:
Incidence of adverse events of pain regimen per Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE version 4.0) | Up to 24 months
  Toxicities will be tabulated by treatment arm using the maximum grade observed by participant. Possible differences by treatment will be described using odds ratio and 95% confidence interval estimates derived use Mantel?Haenszel methods to account for laterality of the radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Anurag Singh, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States